CLINICAL TRIAL: NCT05436704
Title: Is One Pass Enough for the Diagnosis of the Pancreatic Masses During EUS-FNB? A Prospective Study
Brief Title: Is One Pass Enough for the Diagnosis of the Pancreatic Masses During EUS-FNB?
Acronym: ONE PASS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas Mater Domini (Other)
Responsible Party: Sponsor
Other Study IDs: 07-2022
Record Dates: First submitted 2022-06-20; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EUS-FNB
  Interventions: Procedure: EUS-FNB

INTERVENTIONS:
Procedure: EUS-FNB — EUS-FNB

SUMMARY:
Endoscopic ultrasonography (EUS) with tissue acquisition (TA) is nowadays a well-established technique for the sampling of solid lesions pancreatic and non-pancreatic lesions. Major complications after EUS-TA of solid masses are rare. Several studies have been published in the last recent years aimed to identify factors related to a non-diagnostic or false-negative EUS-FNA, and to improve its diagnostic yield using different needle gauge and different tissue acquisition technique as fanning technique, slow-pull stylet extraction or suction technique.

To overcome this problem, new EUS-TA needles entered in clinical practice to obtain histological specimens increasing the accuracy of the EUS-TA. Preliminary result with these new needles, called EUS-fine needle biopsy (FNB) are promising with an accuracy rate more than 90%.

Recently, Leungh et al. conducted an observational study to evaluate the role of macroscopic on-site evaluation (MOSE) on the diagnostic accuracy of 22G Franseen-tip needle. The study demonstrated that MOSE using the 22G Franseen tip needle could limit needle passes by accurately estimating histologic core fragments. However, the study limitations such as the small sample size and the lack of control group, hampered the value of the conclusions.

So, nowadays, no definitive data regarding how many needle passes need to be performed with FNB needles, neither regarding the use of MOSE to evaluate the specimens obtained with FNB needle. The MOSE technique of the acquired tissue was proposed for the first time by Iwashita et al, using a 19G needle and is nowadays a well-established technique with high accuracy in the final diagnosis.

The aim of our study is to evaluate if during EUS-FNB of pancreatic masses only one needle pass with MOSE evaluation can be satisfactory to obtain a correct diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18, both genders.
* Both in-patient and out-patients.
* Presence of a solid lesion. In the presence of a cystic component, the solid part of the lesion should be more 75% of the total.
* FNB performed by a 22G needle Acquire® (Boston Scientific).
* Tissue acquisition with fanning technique.
* Able to obtained informed consent.

Exclusion Criteria:

* Patients underwent EUS-FNA with or without ROSE
* Patients underwent EUS-FNB plus ROSE.
* Previous biopsy of the lesion with diagnosis of malignancy
* Presence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.
* Pregnancy or breast-feeding.
* Patients unable to understand and/or read the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 79 patients with solid pancreatic masses underwent EUS-FNB will be included.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of one pass EUS-FNB. | 24 months
  EUS-FNB only one needle pass inside the target lesions with MOSE evaluation can be satisfactory to obtain a correct diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Mangiavillano, MD, Principal Investigator — benedetto.mangiavillano@mc.humanitas.it
Locations (1):
- Humanitas-Mater Domini, Castellanza, Italy

IPD SHARING:
Plan to Share IPD: No